CLINICAL TRIAL: NCT04443192
Title: A Double-blind, Randomised, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending and Repeated Doses of Orally Administered ZF874 in Healthy Volunteers and PiXZ Subjects
Brief Title: A Single Ascending and Repeated Dose Study of Oral ZF874 in Healthy Volunteers and PiXZ Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the results observed to date, the Sponsor concluded that ZF874 was unlikely to achieve the desired target product profile.
Sponsor: Z Factor Limited (Industry)
Collaborators: Hammersmith Medicines Research (Other); Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZF-0101
Record Dates: First submitted 2020-06-16; First posted 2020-06-23 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Alpha1 Anti-Trypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomised, placebo-controlled, single ascending and repeat dose trial in healthy subjects and subjects carrying at least one Z-A1AT allele (PiXZ subjects)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A Groups 1-6 and Part B Group 1 will be double-blind; Part A Group 7 (food effect) and Part B Groups 2-4 will be open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Part A Cohort 1 - ZF874 (Active Comparator): Single oral dose of ZF874 by mouth in the fasted state. Dose Level 1
  Interventions: Drug: ZF874
- Part A - Placebo to ZF874 - Single Dose (Placebo Comparator): Single oral dose of placebo by mouth in the fasted state
  Interventions: Drug: Placebo
- Part A Cohort 2 - ZF874 (Active Comparator): Single oral dose of ZF874 by mouth in the fasted state. Dose Level 2
  Interventions: Drug: ZF874
- Part A Cohort 3 - ZF874 (Active Comparator): Single oral dose of ZF874 by mouth in the fasted state. Dose Level 3
  Interventions: Drug: ZF874
- Part A Cohort 4 - ZF874 (Active Comparator): Single oral dose of ZF874 by mouth in the fasted state. Dose Level 4
  Interventions: Drug: ZF874
- Part A - Placebo to ZF874 - Two Doses (Placebo Comparator): Two doses of placebo (12 h apart) by mouth in the fasted state
  Interventions: Drug: Placebo
- Part A Cohort 5 - ZF874 - Two Doses (Active Comparator): Two doses of ZF874 (12 h apart) by mouth in the fasted state. Dose Level 5
  Interventions: Drug: ZF874
- Part A Cohort 6 - ZF874 - Two Doses (Active Comparator): Two doses of ZF874 (12 h apart) by mouth in the fasted state. Dose Level 6
  Interventions: Drug: ZF874
- Part A Cohort 7 - ZF874 - Single Dose (Active Comparator): Single oral dose of ZF874 by mouth after consuming a high-fat breakfast. Dose Level 3
  Interventions: Drug: ZF874
- Part B Cohort 1 - ZF874 (Active Comparator): Two doses of ZF874 (12 h apart) by mouth daily for 28 days.
  Interventions: Drug: ZF874
- Part B Cohort 1 - Placebo to ZF874 (Placebo Comparator): Two doses of placebo (12 h apart) by mouth daily for 28 days.
  Interventions: Drug: Placebo
- Part B Cohort 2 - ZF874 (Active Comparator): Two doses of ZF874 (12 h apart) by mouth daily for 28 days.
  Interventions: Drug: ZF874
- Part B Cohort 3 - ZF874 (Active Comparator): Two doses of ZF874 (12 h apart) by mouth daily for 28 days.
  Interventions: Drug: ZF874
- Part B Cohort 4 - ZF874 (Active Comparator): Two doses of ZF874 (12 h apart) by mouth daily for 28 days.
  Interventions: Drug: ZF874

INTERVENTIONS:
Drug: ZF874 — ZF874 is a novel chemical chaperone that is specifically designed to rescue the folding of the Z variant of alpha-1-antitrypsin (A1AT). It is being developed for the treatment of alpha-1-antitrypsin deficiency (AATD) caused by the Z-mutation.
  Arms: Part A Cohort 1 - ZF874; Part A Cohort 2 - ZF874; Part A Cohort 3 - ZF874; Part A Cohort 4 - ZF874; Part A Cohort 5 - ZF874 - Two Doses; Part A Cohort 6 - ZF874 - Two Doses; Part A Cohort 7 - ZF874 - Single Dose; Part B Cohort 1 - ZF874; Part B Cohort 2 - ZF874; Part B Cohort 3 - ZF874; Part B Cohort 4 - ZF874
Drug: Placebo — Placebo to ZF874
  Arms: Part A - Placebo to ZF874 - Single Dose; Part A - Placebo to ZF874 - Two Doses; Part B Cohort 1 - Placebo to ZF874

SUMMARY:
This study is composed of two parts. Part A: will test single doses of ZF874 in a double-blind, randomised, placebo-controlled and dose-escalating design (except Group 7, which will be open-label and without placebo). Up to 7 groups of 6-8 healthy volunteers will receive an oral dose of ZF874 or matching placebo (6 active: 2 placebo in Groups 1-6; 6 active in Group 7). The dosing of the first 2 subjects (1 active and 1 placebo) will take place before dosing of the remainder of the group in Groups 1-6, with morning doses given in the fasted state. The dose will be escalated only if the safety and tolerability of the previous highest dose are acceptable, and the plasma concentrations of ZF874 are predicted to remain below the toxicokinetic exposure limit, as determined by the Safety Review Group. Group 7 will consist of 6 subjects, all of whom will receive ZF874 after consuming a standard high-fat breakfast. Dosing of the first 2 subjects before the rest of the group is not required in Group 7, as 6 subjects have already safely received ZF874 at this dose in Group 3 and 12 subjects have already safely received higher doses in Groups 4 and 5.

The dose selected for Part A, Group 7 was chosen as the dose has previously been given to subjects fasted in Group 3, and it was safe and well tolerated, allowing for comparison for the food effect, and higher doses have been tested in Part A with no safety concerns.

Part B: Multiple Ascending Doses in subjects carrying at least one Z mutated alpha-1-antitrypsin (Z-A1AT) allele (PiXZ subjects): Up to 4 groups of up to 5 PiXZ subjects will be enrolled in Part B (Groups 1-4). In Group 1, up to 4 subjects will receive twice daily doses of either ZF874 or placebo on 28 consecutive days. The dose level (dose and dose regimen) selected for Part B Group 1 will be based on review of the available results from Part A. In Groups 2-4, up to 5 PiXZ subjects will receive ZF874 twice daily by mouth for 28 days; no subjects will receive placebo. The dose for Groups 2 - 4 will not exceed the doses already given in Part A.

DETAILED DESCRIPTION:
Part A: Enrolment of up to 54 healthy men and women is planned, in up to 7 groups. Each of the first 6 groups will consist of 8 subjects and the 7th group will consist of 6 subjects. Subjects will receive either one or two oral dose(s) of either ZF874 or placebo, in the fasted state in the first 6 groups. There will be up to 7 dose levels of ZF874. In each of the first 6 groups, two subjects (one placebo, one ZF874) are to be dosed in a double-blind manner at least 23 hours prior to the remainder of the group. In the absence of any safety concerns in the leading subjects, the remaining subjects will be dosed, at intervals of at least 10 minutes. Dosing of the first 2 subjects before the rest of the group is not required in Group 7, as 6 subjects have already safely received ZF874 at this dose in Cohort 3, and 12 subjects have already safely received higher doses in Cohorts 4 and 5. In Group 7, all subjects will receive a single dose of ZF874 by mouth, after consuming a high-fat breakfast. All subjects will be screened in the 28 days before their dose of trial medication. Subjects will be resident on ward from 1 day before their dose (Day -1) until 48 hours after dosing (Day 3). They will return for a follow-up visit 5-7 days after their dose (Day 6-8).

Part B: In Group 1, up to 4 subjects will receive twice daily doses of either ZF874 or placebo on 28 consecutive days (up to 3 active: up to 2 placebo). The dose level (dose and dose regimen) selected for Part B Group 1 will be based on review of the available results from Part A.

In Groups 2-4, up to 5 PiXZ subjects will receive ZF874 twice daily by mouth for 28 days; no subjects will receive placebo. The doses will be selected after reviewing the available safety and pharmacokinetic results from previous groups, but will not exceed the doses already given in Part A.

Subjects will be pre-screened to confirm PiXZ genotype within 84 days before their dose of trial medication. Once their genotype is confirmed, they will be screened in the 28 days before their dose of study medication. Subjects will be resident on the ward from 1 day before their first dose (Day -1) until 1 hour after they receive their second dose (Day 2). They will then attend 6 outpatient visits before returning to the ward and be resident from Day 27 until 24 hours after the final dose (Day 29). They will return for further outpatient visits on Days 36, 43 and 50, and for a follow-up visit 28-30 days after their final dose (Day 56-58).

ELIGIBILITY:
Inclusion Criteria:

* Part A: healthy Caucasian males or females, aged 18-65 years at the time of consent; Part B: males or females of general good health, aged 18-72 years at the time of consent.
* Body mass index of 18.0-30.0 kg/m^2 (Part A) and 18.0-35.0 kg/m^2 (Part B).
* Able to understand the nature of the trial and any hazards of participating in it. Able to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of the entire trial
* Willing to give written fully informed consent to participate
* Agree to follow the contraception requirements of the trial
* Agree not to donate blood or blood products during the study and for up to 3 months after the trial medication
* Registered with a General Practitioner in the United Kingdom
* Willing to give written consent to have data entered into The Over-volunteering Prevention System [Part B only]
* Confirmed genotype with at least one Z alpha-1-antitrypsin allele (PiXZ)

Exclusion Criteria:

* Woman who is pregnant or lactating, or woman of child-bearing potential who is sexually active and not using a highly effective method of contraception
* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer
* Acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness
* Creatinine clearance <60 mL/min/1.73m2
* Active cancer or to be actively on cancer therapy, or diagnosis of cancer (except for Basal Cell Carcinoma, Squamous Cell Carcinoma (fully excised), or Cervical Intra-epithelial Neoplasia in situ) in the 5 years before the first dose of trial medication.
* Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines
* Presence or history of severe adverse reaction to any relevant drug
* During the 28 days before the first dose of trial medication, the use of prescription medicine judged by the investigator to have the potential to influence the results of the study; or during the 7 days before the first dose of trial medication, the use of a herbal supplement or an over-the-counter medicine, with the exception of ibuprofen
* Receipt of a COVID-19 vaccine within 14 days before the first dose of trial medication; exhibition of symptoms suspected to be related to COVID-19 within 28 days before the first dose of trial medication; or receipt of a positive COVID-19 test during the 28 days before the first dose of trial medication
* Receipt of an investigational product (including prescription medicines) as part of another clinical trial within 3 months before admission to this study; in the follow-up period of another clinical trial at the time of screening for this study
* Recent drug or alcohol abuse (within 2 years before screening), or intake of more than 3 units of alcohol daily (for men) or 2 units of alcohol daily (for women); or use of cigarettes or nicotine-containing products during 30 days before the first dose of trial medication until the end of the study
* Blood pressure and heart rate in supine position at the screening examination outside the ranges: blood pressure 90-160 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40-100 beats/min
* Possibility that the volunteer will not cooperate with the requirements of the protocol
* Evidence of drug abuse on urine testing
* Positive test for hepatitis B virus, hepatitis C virus or human immunodeficiency virus
* Loss of more than 400 mL blood during 3 months before the trial, eg as a blood donor
* Objection by General Practitioner to volunteer entering trial

Part A, Cohort 7 only:

- Vegans, vegetarians, or unwilling to eat a high-fat breakfast containing bacon.

Part B only:

- Undergone liver transplantation

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | Part A: Day 1 to Day 8; Part B: Day 1 to Day 58
  Safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part A: Day 1 to Day 3; Part B: Day 1 to Day 29
  maximum plasma concentration
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part A: Day 1 to Day 3; Part B: Day 1 to Day 29
  time of maximum plasma concentration
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part B: Day 1 to Day 29
  trough plasma concentration
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part A: Day 1 to Day 3; Part B: Day 1 to Day 29
  maximum plasma concentration / dose
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part A: Day 1 to Day 2
  area under the concentration-time curve during the 24 hours post-dose area under curve to 24 hours post-dose
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part A: Day 1 to Day 3
  area under the concentration-time curve during the 48 hours post-dose area under the concentration-time curve to 48 hours post-dose
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part B: Day 1 to Day 29
  area under the concentration-time curve during the dosing interval
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part A: Day 1 to Day 3; Part B: Day 1 to Day 29
  area under the concentration-time curve to last measurable concentration
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part A: Day 1; Part B: Day 28
  terminal elimination half-life
Pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects and PiXZ subjects | Part A: Day 1; Part B: Day 28
  terminal rate constant
Food effect on the pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects | Part A: Day 1 to Day 3
  maximum plasma concentration / dose
Food effect on the pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects | Part A: Day 1 to Day 3
  area under the concentration-time curve to last measurable concentration
Food effect on the pharmacokinetics of ZF874 and its metabolite ZF857 in healthy subjects | Part A: Day 1 to Day 3
  area under the concentration-time curve extrapolated to infinite time

OTHER OUTCOMES:
Pharmacodynamics (Exploratory) | Part B: Day 1 to Day 58
  Serum levels of Z-mutated alpha-1-antitrypsin (Z-A1AT)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, BSc MD FRCP FFPM, Principal Investigator — HMR; Giuseppe Fiore, MSc MD, Principal Investigator — MAC Clinical Research
Locations (5):
- United Kingdom (5):
  - MAC Clinical Research Manchester, Manchester, Greater Manchester
  - MAC Clinical Research, Barnsley, Barnsley
  - MAC Clinical Research, Leeds, Leeds
  - Hammersmith Medicines Research, London
  - MAC Clinical Research, Teesside, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No